CLINICAL TRIAL: NCT01081067
Title: Assessment of Efficiency and Safety of an Infant Formula Containing a Probiotic in Children
Status: Completed | Type: Observational
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Deolinda Scalabrin, M.D., Mead Johnson Nutrition
Other Study IDs: 3377-1 (6008)
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Stool Output

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Routine cow milk-based infant formula
- Investigational: Cow milk-based infant formula containing probiotics

SUMMARY:
Evaluate the effect of probiotics on stool output in children 1 - 18 months old.

DETAILED DESCRIPTION:
Evaluate the effect of probiotics on stool output in children 1 - 18 months old.

ELIGIBILITY:
Inclusion Criteria:

* children 1 - 18 months of age
* acute diarrhea
* adequately hydrated
* signed informed consent

Exclusion Criteria:

* exclusively or predominantly breast-feeding
* bloody diarrhea
* intercurrent illnesses that may affect study parameters
* use of systemic antibiotics during the 72 hours prior to enrollment
* use of anti-diarrheal medications at the time of enrollment
* use of supplement or infant formula with Lactobacillus rhamnosus 10 days prior to enrollment

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: CPPHO [Centro Pediátrico Professor Hosannah de Oliveira (Professor Hosannah de Oliveira Pediatirc Center] C-HUPES [Complexo Hospitalar Professor Edgar Santos (Professor Edgar Santos Hospital Complex)]
Sampling Method: Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Ribeiro, Jr., M.D., Principal Investigator — Professor Edgard Santos University Hospital - UFBA
Locations (1):
- Metabolic Unit Fima Lifshitz, Federal University of Bahia School of Medicine, Salvador, Estado de Bahia, Brazil